CLINICAL TRIAL: NCT00842907
Title: A Clinical, Laboratorial and Quality of Life Study to Evaluate the Efficacy and Safety of Oral Isotretinoin in the Treatment of Cutaneous Photodamage
Brief Title: Efficacy and Safety of Oral Isotretinoin for Cutaneous Photodamage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Edileia Bagatin, MD, PhD, Federal University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNICCO
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2009-04

CONDITIONS: Photodamage; Photoaging
Keywords: Brazil; isotretinoin; photodamage; photoaging
MeSH Terms: interventions — Isotretinoin; Retinoids; Tretinoin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral isotretinoin (Active Comparator): Twelve subjects will be treated with oral isotretinoin 20.0 mg, once a day, every other day, for 24 weeks.
  Interventions: Drug: oral isotretinoin
- tretinoin (Active Comparator): Twelve patients will be treated with 0,05% tretinoin cream applied on face and forearms at night and moisturizer broad-spectrum sunscreen twice a day.
  Interventions: Drug: Tretinoin

INTERVENTIONS:
Drug: oral isotretinoin — one 20.0 mg capsule, once a day, every other day, during 24 weeks
  Other Names: oral retinoid
  Arms: oral isotretinoin
Drug: Tretinoin — 0.05% tretinoin cream applied on face and forearms, once a day, in the night, during 24 weeks
  Other Names: topical retinoid; topical tretinoin; topical retinoic acid
  Arms: tretinoin

SUMMARY:
This is a randomized, comparative, single evaluator-blinded trial to evaluate clinical, histological and immunohistochemical effects of oral isotretinoin plus moisturizer sunscreen as compared to the use of 0,05% tretinoin cream plus moisturizer sunscreen for the treatment of photodamage on face and forearms. Main oral isotretinoin safety parameters will also be analyzed, as well as adverse events related to topical products.

DETAILED DESCRIPTION:
A 24-week study, with 7 or 9 monthly visits, comprising healthy adult volunteers, aged 50 to 75 years will be carried out. The patients should present advanced to severe photodamage on face and forearms. Written informed consent will be obtained from each subject prior to enrollment.

Eligible patients will be randomly divided in two groups:

A- 10 patients will be treated with oral isotretinoin, 20.0 mg/day, every other day, 15 capsules per month, for 24 weeks, associated with the use of moisturizer broad spectrum sunscreen twice a day.

B- 10 patients (controls) will be treated with 0,05% tretinoin cream applied on face and forearms at night and the same moisturizer broad-spectrum sunscreen twice a day.

After randomization, laboratory tests will be requested for patients from group A and will be repeated on weeks 4 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 50 to 75 years old
* Post-menopausal women for at least one year
* Patients with moderate to severe photodamage on face and arms
* Individuals in generally good health
* Fitzpatrick I to III skin type
* Patients who are willing to avoid sun-exposure during the study period

Exclusion Criteria:

* Patients of child bearing potential
* Individuals who have been treated with topical anti-aging products and/or superficial chemical peels within 3 months or received topical tretinoin or oral retinoid (6 months); fillers and/or botulinum toxin applications (4 months); medium-depth chemical peels or ablative lasers or dermabrasion (6 months) and surgical lifting (12 months) will not be eligible for inclusion in the study
* Patients on cytotoxic drugs (including azathioprine, cyclophosphamide, mycophenolate mofetil, or other chemotherapeutic agents) within 3 months
* Hypersensitivity to parabens
* An infectious or inflammatory dermatosis of the face, scalp or forearms including acne rosacea
* A history of photodermatosis (example PMLE)
* Immunocompromised individuals
* Patients with auto-immune diseases
* Patients addicted to drugs or alcohol

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-12 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Clinical, histological and immunohistochemical features before and after treatments | 24 weeks

SECONDARY OUTCOMES:
Quality of life | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edileia Bagatin, MD, PhD, Principal Investigator — Federal University of Sao Paulo, Brazil
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil